CLINICAL TRIAL: NCT00199238
Title: A 4-week Dose-finding, Multicentre, Double-blind, Randomised, Placebo-controlled, Parallel-group Trial to Assess the Efficacy and Safety of Different Doses of Rupatadine Compared to Placebo in the Treatment of Chronic Idiopathic Urticaria
Brief Title: Efficacy of Rupatadine 5, 10 and 20 mg in Chronic Idiopathic Urticaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: J. Uriach and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002/47
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: URTICARIA
Keywords: ANTIHISTAMINE; RUPATADINE; WHEAL; FLARE; DERMATOLOGY
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Once daily/ 28 days
  Interventions: Drug: Rupatadine Fumarate
- rupatadine 5mg (Experimental): Once daily/ 28 days
  Interventions: Drug: Rupatadine Fumarate
- rupatadine 10 mg (Experimental): Once daily/ 28 days
  Interventions: Drug: Rupatadine Fumarate
- rupatadine 20 mg (Experimental): Once daily/ 28 days
  Interventions: Drug: Rupatadine Fumarate

INTERVENTIONS:
Drug: Rupatadine Fumarate
  Other Names: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of rupatadine for the treatment of CIU symptoms.To assess the clinical efficacy of a dose ranging of rupatadine fumarate (5mg, 10mg, and 20 mg) compared with placebo for relief of CIU symptoms.

DETAILED DESCRIPTION:
Objectives: To evaluate the efficacy and safety of rupatadine for the treatment of CIU symptoms.To assess the clinical efficacy of a dose ranging of rupatadine fumarate (5mg, 10mg, and 20 mg) compared with placebo for relief of CIU symptoms.

Methodology: A dose-finding multicentre, double-blind, randomised, placebo-controlled, parallel-group study Number of patients (planned and analysed): 248 patients. 62 patients will be allocated to each treatment group. 283 patients were randomised and analysed.

Diagnosis and criteria for inclusion: Man or woman aged between 12 and 65. Documented history of active CIU (urticaria wheals) with or without an associated angioedema for at least three days per week over the last 6 weeks prior to Day 0 . Active CIU (score ³2 labelled as moderate pruritus) for at least 3 days (not necessarily consecutive days) in the week before inclusion with a total score of active CIU ³6 labelled as moderate pruritus for these 3 days. Results of standard laboratory biochemistry and haematology tests obtained at screening within acceptable limits as assessed by investigator. Patient who signed the informed consent form.

Test product, dose, mode of administration, batch N°: Rupatadine 5,10 and 20 mg tablets; oral dose of 1 tablet/day for 4 consecutive weeks; batch 0102 (France) and batch 0203 (Hungary, Romania and Argentina). Expiry date: 12/2003 (France) and 10/2004 (Hungary, Romania and Argentina).

Duration of treatment: Oral administration of test formulation (5, 10, 20 mg) or placebo daily, for 4 consecutive weeks.

Reference therapy: Placebo tablets, 1 tablet/day for 4 consecutive weeks. Criteria for evaluation (efficacy): Primary efficacy measure of each treatment will compare the frequency and severity of symptoms of CIU as measured by the patient in terms of change in mean pruritus score (MPS) over the 4-week treatment period.Secondary efficacy measures include change from baseline over the 4-week treatment period in the mean number of wheals (MNW) score; mean total symptoms score (MTSS), calculated as the sum of the MPS (Mean pruritus symptoms) and the MNW (Mean number of wheals) scores and the interference with sleep and daily activities due to urticaria symptoms Criteria for evaluation (safety): AEs, laboratory tests and vital signs

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged between 12 and 65
2. Documented history of active CIU (urticaria wheals) with or without an associated angioedema for at least three days per week over the last 6 weeks prior to Day 0
3. Active CIU (score ³2 labelled as moderate pruritus) for at least 3 days (not necessarily consecutive days) in the week before inclusion with a total score of active CIU ³6 labelled as moderate pruritus for these 3 days
4. Results of standard laboratory biochemistry and haematology tests obtained at screening within acceptable limits as assessed by investigator
5. Patient who signed the informed consent form -

Exclusion Criteria:

1. CIU associated to some underlying disease (Hodgkin's disease/vasculitis/lupus erythematous/hepatitis)
2. Patient under any systemic or topical medication for CIU and/or an inferior wash-out period as stated as follows:

   * H1-receptor antagonists: fexofenadine (10 days prior to Day 0), loratadine, cetirizine, hydroxyzine, diphenhydramine, cyproheptadine, etc. (3 days prior to Day 0)
   * H2-receptor antagonists: cimetidine, ranitidine and famotidine (2 days prior to Day 0)
   * H1- and H2-receptor antagonists: doxepin (7 days prior to Day 0)
   * Leukotriene antagonists: zafirlukast and montelukast (4 days prior to Day 0)
   * Corticosteroids: prednisone and methylprednisolone (7 days prior to Day 0)
   * Tricyclic antidepressants: imipramin and amitriptilin (30 days prior to Day 0)

   The informed consent form must be signed prior to any washout period is set up.
3. Physical urticaria due to cold, heat, and/or sun
4. Cholinergic urticaria
5. Patient taking any potential inhibitors of the CYP3A4 isozyme of cytochrome P450 such as ketoconazole, erythromycin and/or tricyclic antidepressants, e.g. imipramin, amitriptilin, etc.
6. Urticaria due to known aetiology (e.g., medications, insects bites, food, etc)
7. Patient unresponsive to antihistaminic treatment
8. Patient with psychiatric disorders, vascular, hepatic, neurological, endocrine or other major systemic disease
9. Pregnant or lactating female
10. Patient with any heart abnormality of clinical relevance or any pathological changes of the heart rate
11. Patient under any medication which could interfere with drug effect or with interpretation of efficacy parameters
12. Subject handling dangerous machinery or driving as an integral part of his/her occupation
13. Patient with hereditary angioedema or isolated dermographism
14. Patient with disease caused by a parasite

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2002-10-28 (Actual); Primary Completion 2003-11-25 (Actual); Study Completion 2004-09-27 (Actual)

PRIMARY OUTCOMES:
Pruritus | 4 weeks
  change in mean pruritus score (MPS) over the 4-week treatment period.

SECONDARY OUTCOMES:
Wheals | 4 weeks
  change in mean number of wheals score (MNW) over the 4-week treatment period.
change in mean total symptoms score (MTSS) over the 4-week treatment period. | 4 weeks
overall impression | 4 weeks
  overall impression for efficacy was done by the investigator and by the patient

CONTACTS AND LOCATIONS:
Overall Officials: EVA Arnaiz, PhD, Study Director — J. Uriach y Compañía
Locations (1):
- Hospital Saint Louis, Paris, France

REFERENCES:
- [Result] Dubertret L, Zalupca L, Cristodoulo T, Benea V, Medina I, Fantin S, Lahfa M, Perez I, Izquierdo I, Arnaiz E. Once-daily rupatadine improves the symptoms of chronic idiopathic urticaria: a randomised, double-blind, placebo-controlled study. Eur J Dermatol. 2007 May-Jun;17(3):223-8. doi: 10.1684/ejd.2007.0153. Epub 2007 May 4. PMID 17478385